CLINICAL TRIAL: NCT00447525
Title: Comparison of the Immunogenicity and Safety of a Combined Adsorbed Low Dose Diphtheria, Tetanus and Inactivated Poliomyelitis Vaccine (REVAXIS®) With a Combined Diphtheria, Tetanus and Inactivated Poliomyelitis Vaccine (DT Polio®) When Given as a Booster Dose at 6 Years of Age
Brief Title: REVAXIS® Versus DT Polio® as a Second Booster in 6 Year-old Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F05-TdI-301
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diphtheria; Tetanus; Poliomyelitis
Keywords: Prevention of : Diphtheria, Tetanus and Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: REVAXIS®
- 2 (Active Comparator)
  Interventions: Biological: DT-Polio®

INTERVENTIONS:
Biological: REVAXIS®
  Arms: 1
Biological: DT-Polio®
  Arms: 2

SUMMARY:
Primary objective:

To demonstrate the non inferiority between REVAXIS® and DT Polio® when given as a second booster to healthy 6 year-old children .

Secondary objectives:

* Additional immunogenicity assessments.
* To describe the safety profile of a single dose of REVAXIS® or DT-Polio®

ELIGIBILITY:
Inclusion Criteria:

1. Healthy child without chronic severe disease of either gender,
2. 6 year-old child on vaccination day,
3. Child previously vaccinated with three doses of a diphtheria, tetanus and poliomyelitis containing vaccine given alone or in combination within the first 6 months of life and a booster dose of a diphtheria, tetanus and poliomyelitis containing vaccine given alone or in combination at 16 - 18 months of life (±2 months),
4. Consent form signed by both parents, or by the legal representative, properly informed about the study.

Exclusion Criteria:

1. Child who had received less or more than 4 doses of a diphtheria, tetanus and/or poliomyelitis containing vaccine,
2. Previous clinical or bacteriological diagnosis of diphtheria, tetanus or poliomyelitis,
3. Child who had received any vaccine in the previous 30 days or with a vaccination scheduled during the course of the study,
4. Child who present with immune impairment or humoral/cellular deficiency, neoplastic disease or depressed immunity,
5. Child who had received within the previous 150 days or who will receive during the course of the study, any immunoglobulins or blood derived products,
6. Child with true hypersensitivity to at least one of the components of a study vaccine or to streptomycin, neomycin or polymixin B,
7. Known personal history of encephalopathy, seizure disorder or progressive, evolving or unstable neurological condition,
8. Child who had presented severe hypersensitivity following an earlier immunization against diphtheria and/or tetanus,
9. Known history of thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection,
10. Acute severe febrile illness and/or oral temperature ≥37.5°C at the time of vaccination

Ages: 6 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 760 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (62):
- France (62):
  - Albertville
  - Albi
  - Angers
  - Annecy
  - Anzin
  - Arras
  - Asnières
  - Avion
  - Bassens
  - Bersée
  - Besançon
  - Blois
  - Boulogne
  - Brest
  - Broglie
  - Caen
  - Chalon-en-champagne
  - Champdeniers
  - Chigny-les-Roses
  - Cholet
  - Claix
  - Clamart
  - Collombey Les Belles
  - Draguignan
  - Enghien-les-Bains
  - Floirac
  - Frouard
  - Haguenau
  - Illkirch-Graffenstaden
  - Issy-les-Moulineaux
  - La Neuville-Roy
  - Laon
  - Le Havre
  - Les Pieux
  - Louverné
  - Louvigné-de-Bais
  - Manduel
  - Marcq-en-barouel
  - Maromme
  - Marseille
  - Miniac-Morvan
  - Montpellier
  - Montsang/orge
  - Morangis
  - Nancy
  - Nantes
  - Nogent-sur-Marne
  - Ostwald
  - Paris
  - Plouzané
  - Poitiers
  - Pont-à-Mousson
  - Quimper
  - Rouen
  - Saint Sebastien Sur Loir
  - Saint-Ouen
  - Saint-Raphaël
  - Sanary Mer
  - Sèvres
  - Strasbourg
  - Toulouse
  - Villemomble

REFERENCES:
- [Derived] Gajdos V, Soubeyrand B, Vidor E, Richard P, Boyer J, Sadorge C, Fiquet A. Immunogenicity and safety of combined adsorbed low-dose diphtheria, tetanus and inactivated poliovirus vaccine (REVAXIS ((R))) versus combined diphtheria, tetanus and inactivated poliovirus vaccine (DT Polio ((R))) given as a booster dose at 6 years of age. Hum Vaccin. 2011 May;7(5):549-56. doi: 10.4161/hv.7.5.14982. Epub 2011 May 1. PMID 21441781